CLINICAL TRIAL: NCT00114842
Title: MR Colonography With Fecal Tagging: A Prospective, Randomized Study
Brief Title: Magnetic Resonance (MR) Colonography With Fecal Tagging
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Herlev Hospital (Other)
Collaborators: University Hospital, Gentofte, Copenhagen (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: KA05029-MA; KA05029
Record Dates: First submitted 2005-06-17; First posted 2005-06-20 (Estimated); Last update posted 2007-09-20 (Estimated); Status verified 2007-09

CONDITIONS: Colorectal Cancer; Polyps
Keywords: colorectal polyps; colorectal cancer; Virtual colonoscopy; Fecal tagging; MR colonography
MeSH Terms: conditions — Colorectal Neoplasms; Polyps

INTERVENTIONS:
Procedure: MR colonography

SUMMARY:
The purpose of this study is to determine if MR colonography with fecal tagging is better using air or water for distension of the colon. Patients referred to colonoscopy are offered MR colonography before colonoscopy. Two days before colonography, patients ingest a 200 ml Barium sulfate solution 2% four times a day, which will render fecal masses "invisible" on the following MR colonography. Air or water (randomised trial) is used for distension of the colon. The examinations are evaluated by two independent blinded readers.

ELIGIBILITY:
Inclusion Criteria:

* Suspicion of colorectal polyps or cancer
* Referred for colonoscopy

Exclusion Criteria:

* Suspicion of IBD
* Pacemaker
* Metal in the body
* Claustrophobia
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2006-03; Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Sensitivity/specificity for water versus air for distension of colon in MR colonography

SECONDARY OUTCOMES:
Feasibility of MR colonography with fecal tagging
Sensitivity/specificity of MR colonography versus colonoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Michael P Achiam, M.D., Principal Investigator — Department of Radiology Copenhagen University Hospital Herlev
Locations (1):
- Department of Radiology Copenhagen University Hospital Herlev, Herlev, Denmark